CLINICAL TRIAL: NCT00489723
Title: Is There is a Role of Prophylactic Therapy With Tamsulosin Before Extracorporeal Shock Wave Lithotripsy to Avoid Development of Steinstrasse ?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Other Study IDs: 0056-07-EMC
Record Dates: First submitted 2007-06-19; First posted 2007-06-21 (Estimated); Last update posted 2007-06-21 (Estimated); Status verified 2007-06

CONDITIONS: Kidney Stones
Keywords: size of stone 1-2 cm; Pt. with no use of alfa bloker prior ESWL; Pt. without internal stent
MeSH Terms: conditions — Kidney Calculi | interventions — Tamsulosin

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: tamsulosin 0.4mg

SUMMARY:
The purpose of this study is to determine if there is a role of prophylactic therapy with tamsulosin prior extracorporeal shock wave lithotripsy to avoid development of steinstrasse. 150 persons that will go to Extracorporeal shock wave lithotripsy will randomize to 2 groups.

Group 1 -of 75 persons will recieve tamsulosin 0.4 mg x 1/d 2 days before the lithotripsy .

Group 2 - of 75 persons will not recieve tamsulosin. 48 hour after the ESWL all 2 group will take abdominal radiograph to evaluate the presence of steinstrasse.

ELIGIBILITY:
Inclusion Criteria:

* size of stone 1-2 cm

Exclusion Criteria:

* ureteral stricture Presence of internal stent prior use of alfa bloker prior ESWL

Ages: 15 Years to 85 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2007-05

CONTACTS AND LOCATIONS:
Overall Officials: doron perez, Principal Investigator — Urology department: Haemek Medical Center
Locations (1):
- Haemek medical center, Afula, Israel